CLINICAL TRIAL: NCT04165174
Title: A Single Arm, Observational Clinical Trial to Evaluate the Efficacy and Safety of Combination Treatment With PD-1 Monoclonal Antibody Plus Apatinib and SBRT in HCC With PVTT
Brief Title: PD-1 Monoclonal Antibody Plus Apatinib Combined With SBRT in HCC With PVTT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Head of the cancer center, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJCC 010
Record Dates: First submitted 2019-10-01; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: HCC
Keywords: HCC; PVTT; PD-1; Apatinib; SBRT
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PAS (Experimental): PD-1:240mg,ivdrip,Q3W,begin with SBRT Apatinib:250mg,po,QD,begin with SBRT SBRT:6-10Gy/F,5-8F
  Interventions: Drug: Terepril monoclonal antibody; Apatinib; Radiation: SBRT

INTERVENTIONS:
Drug: Terepril monoclonal antibody; Apatinib — Terepril monoclonal antibody,240mg,ivdrip,Q3W Apatinib,250mg,po,QD
Radiation: SBRT — 6-10Gy/F,5-8F

SUMMARY:
It is a trial to assess the efficacy and safety of PD-1 monoclonal antibody plus Apatinib combined with SBRT as first-line treatment in HCC with PVTT.

ELIGIBILITY:
Inclusion Criteria:1. Age of 18-75 years old;

2. Patients with primary hepatocellular carcinoma confirmed by cell or histopathology were complicated with PVTT and BCLC stage C.

3. According to RECIST criteria, there is at least one measurable lesion, which is a lesion other than SBRT.

4. Child-Pugh A or partial B grade of liver function (recovered to A grade after supportive treatment); normal liver volume > 700 ml;

5. Renal function: Serum creatinine < 1.5 times normal upper limit;

6. ECOG score 0-1;

7. The life expectancy is more than 3 months.

8. There were no obvious signs of hematological diseases, ANC (> 1.5 *109/L), platelet count (> 75 *109/L) and no tendency of bleeding before enrollment, HGB (> 90 g/L) and INR (< 2.5 times normal upper limit and APT (< 1.5 times normal upper limit).

9. FT3, FT4 and TSH are within the normal range of 10%.

10. No history of abdominal irradiation.

11. Patients with other previous malignant tumors had a disease-free survival of more than 2 years after initial treatment (e.g. non-melanoma skin cancer or cervical cancer in situ).

12. The patient signed the informed consent.

13. Female patients of childbearing age or male patients whose sexual partners are women of childbearing age need to take effective contraceptive measures during the whole treatment period and within 6 months after treatment.

14.It is better to provide tissue samples for biomarker analysis (e.g. PD-L1) and to optimize newly acquired tissues. Patients who are unable to provide newly acquired tissues can provide 5-8 paraffin sections of 3-5 micron thickness for archival preservation.

-

Exclusion Criteria:1. Fibrous layer hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma and mixed hepatocellular carcinoma;

2. History of hepatic encephalopathy or liver transplantation;

3. Pleural effusion, ascites and pericardial effusion with clinical symptoms or needing drainage. Only a small amount of pleural effusion, ascites and pericardial effusion, asymptomatic;

4. Untreated hepatitis infection: HBV DNA > 2000iu/ml, HCV RNA > 103copy/ml, HBsAg and anti-HCV antibodies were positive.

5. Distant metastasis.

6. In the past six months, there have been history of gastrointestinal perforation and/or fistula, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), inflammatory bowel disease or extensive intestinal resection (partial or extensive enterectomy for chronic diarrhea), Crohn's disease, ulcer, etc. Acute colitis or chronic diarrhea;

7. Symptomatic history of interstitial lung disease or other conditions that may lead to confusion in the detection or management of suspected drug-related pulmonary toxicity;

8. Evidence of active pulmonary tuberculosis (TB). Patients diagnosed with active pulmonary tuberculosis infection within one year should be excluded even if they have received treatment.

9. Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS) positive;

10. Severe infections are active or under clinical control. Severe infections occurred within 4 weeks before the first treatment, including but not limited to hospitalization due to infections, bacteremia or complications of severe pneumonia.

11. Patients with active, known or suspected autoimmune diseases. Patients with vitiligo, type I diabetes mellitus, thyroid dysfunction caused by autoimmune thyroiditis (only hormone replacement therapy) or diseases that do not recur without external stimuli can be selected.

12. Immunosuppressive drugs used in the past four weeks, excluding local or systemic glucocorticoids (i.e., prednisone or other equivalent doses of glucocorticoids not exceeding 10 mg/day), through nasal sprays, inhalation or other routes, and temporarily using glucocorticoids to treat dyspnea symptoms of asthma, Chronic obstructive pulmonary disease;

13. Any anti-infective vaccines (such as influenza vaccine, varicella vaccine, etc.) have been vaccinated in the past four weeks.

14. Receiving systemic immune stimulation therapy in the past four weeks;

15. In the past four weeks, major operations (craniotomy, thoracotomy or laparotomy) or unhealed wounds, ulcers or fractures have been performed.

Uncontrolled metabolic disorders or other non-malignant organs or systemic diseases or secondary tumors may lead to higher medical risks and/or uncertainty in survival assessment;

17. Laboratory test values for some acute or chronic diseases, psychiatric disorders or abnormalities that may lead to outcomes: increased risk of participating in research or drug management, or interference with the interpretation of research results, according to the judgement of researchers, patients are classified as not eligible to participate in research;

18. Other malignant tumors were diagnosed within five years before the first administration, excluding cured basal cell carcinoma of the skin, cured squamous cell carcinoma and/or in situ cured cancer. If other malignant tumors or hepatocellular carcinomas are diagnosed more than 5 years before administration, pathological or cytological diagnosis should be made from the sites of recurrence and metastasis.

19. Use anti-PD-1/PD-L1/PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell co-stimulation or checkpoint pathway) for any prior immunosuppressive treatment.

20. Patients with known sensitivity or allergy to any component of humanized anti-PD-1 antibody or Apatinib;

21. Pregnancy and breastfeeding.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 3 years
  PFS is defined as time from the start of treatment to progression of disease or death.

SECONDARY OUTCOMES:
OS | up to 3 years
  Overall survival is defined as time from the start of treatment until death due to any reason.
ORR | up to 3 years
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
DCR | up to 3 years
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
TTSP | up to 3 years
  The time between the onset of randomized grouping and the onset of symptomatic progression.
Safety as measured by number and grade of adverse events | up to 3 years
  Summary adverse events according to NCI-CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, MD,PhD, Study Chair — Tongji Hospital
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China